CLINICAL TRIAL: NCT06222970
Title: Maxillary Sinus Augmentation Via the "Bone Lid Technique"
Acronym: SINUSLID_2023
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Antonio Barone, Full Professor of Oral Surgery and Implantology, Principal Investigator, University of Pisa
Other Study IDs: SINUSLID_2023
Record Dates: First submitted 2024-01-15; First posted 2024-01-25 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Maxillary Deficiency
MeSH Terms: conditions — Retrognathia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bone lid repositioning in course of sinus lift — A full-thickness flap was elevated to access the lateral maxillary bone wall. Subsequently, a lateral access window was prepared using a piezoelectric device with specific bone tips, delimitating a trapezoidal bone lid.
  Once the antrostomy was completed, the bone lid was gently removed with a Lucas surgical curette and anatomical tweezers, with great care to avoid damages to the Schneiderian membrane. The Schneiderian membrane was detached from the bone layer using specific sinus curettes. In case of sinus membrane perforation, the membrane was raised in all directions. All clinical cases received a cortical bone lamina to avoid graft particles displacement in the maxillary sinus. The elevated space was filled with chips of cortico-spongious bone. The antrostomy was then covered with the bone lid (osteotomy window), previously removed and preserved in physiological solution and fixed in the original anatomical position with a surgical glue. The flap was then repositioned and sutured.

SUMMARY:
Maxillary sinus augmentation is one of the most performed procedures to increase the bone quantity of the atrophic maxilla in order to allow implant placement. The aim of the present case series was to describe a surgical protocol to perform maxillary sinus augmentation with the "bone lid technique", and its outcomes in a cohort of patients eligible for the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Partially or fully edentulous patients requiring an implant-prosthetic rehabilitation of the premolar or molar maxillary areas with a residual ridge height lower than 4 mm.
* Patients needing for a unilateral or bilateral sinus lift with a lateral wall approach.

Exclusion Criteria:

* Patients under treatment with immunosuppressive agents
* Patients under treatment with medications that could impair bone metabolism.
* Patients pregnant or breastfeeding.
* Patients who had received irradiation treatment to the head and neck area.
* Patients with uncontrolled diabetes.
* Patients with uncontrolled periodontal disease.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients referred to the Unit of Dentistry and Oral Surgery, University Hospital of Pisa, with a severe bone atrophy of the maxillary posterior areas that required bone grafting through a lateral approach of the maxillary sinus
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-05-04 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Bone gain | 6 months
  Measurement of bone height and width

CONTACTS AND LOCATIONS:
Locations (1):
- U.O. Odontostomatologia e Chirurgia del Cavo Orale, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No
data will be published after anonymization and/or as aggregated data